CLINICAL TRIAL: NCT04028531
Title: Understanding Chronic Lymphocytic Leukemia
Status: Recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer R. Brown, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 99-224; R01CA213442-01A1 (NIH)
Record Dates: First submitted 2019-06-26; First posted 2019-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — peripheral blood mononuclear cells, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sample Collection: * Blood tests required for assessment
  * Specimens and data will also be collected from outside sites
  * Clinical data from patients with Chronic Lymphocytic Leukemia will be gathered into a database at Dana Farber Cancer Institute

SUMMARY:
The purpose of this study is to collect human Chronic Lymphocytic Leukemia tissue samples and medical information, in order to find out more about the causes and biology of chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
The purpose of this study is to collect human Chronic Lymphocytic Leukemia tissue samples and medical information, in order to find out more about the causes and biology of chronic lymphocytic leukemia, for the potential development of more effective therapies for this disease.

ELIGIBILITY:
Inclusion Criteria:

* New and existing patients seen for treatment of monoclonal B-cell lymphocytosis
* Any low grade lymphoproliferative disorder
* Chronic Lymphocytic Leukemia in the Dana Farber Cancer Institute Hematologic Oncology Clinic or elsewhere

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Monoclonal B-cell lymphocytosis or Chronic Lymphocytic Leukemia in any phase of their disease.
Sampling Method: Non-Probability Sample
Enrollment: 2750 (Estimated)
Dates: Start 1999-09-29 (Actual); Primary Completion 2030-09-29 (Estimated); Study Completion 2032-09-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of novel genomic prognostic markers in Chronic Lymphocytic Leukemia | 20 years
  Exploratory science to better understand Chronic Lymphocytic Leukemia

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brown, MD,PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Boston Childrens Hospital - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu Brigham and Women's Hospital - Contact the Partners Innovations team at http://www.partners.org/innovation Dana Farber Cancer Institute - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu Massachusetts General Hospital - Contact the Partners Innovations team at http://www.partners.org/innovation